CLINICAL TRIAL: NCT05814055
Title: The Potential of Kava in Enabling Tobacco Cessation - Its Holistic Effects in Managing Stress and Insomnia Associated With Abstinence
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Kava 2; OCR44061 (Other: University of Florida); IRB202300887 (Other: University of Florida); 1R33AT012328-01 (NIH)
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Smoking
Keywords: kava; smoking cessation; tobacco dependence
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AB-free kava (Experimental)
  Interventions: Drug: AB-free kava
- Placebo control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Participants on this arm will take one placebo capsule orally three times daily for 4 weeks.
  Arms: Placebo control
Drug: AB-free kava — Participants on this arm will take one kava capsule (each capsule contains 75 mg of kavalactones) orally three times daily for 4 weeks.
  Arms: AB-free kava

SUMMARY:
This study will evaluate the compliance with a daily kava regimen among active smokers who have an intention to quit smoking. This study will also investigate whether kava use can facilitate tobacco cessation, reduce stress, and improve sleep.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 21 years or above (legal age for smoking in the U.S.) up to 75 years old;
* self-reported smoking at least 5 cigarettes/day for the past year with INTENTION to quit at time of screening visit;
* expired carbon monoxide level of more than 8 ppm at recruitment;
* willingness to participate in the proposed study, as indicated by signed informed consent;
* access to a functional telephone;
* expected presence in the study's geographical area for the next 4 months;
* not currently enrolled in any smoking cessation programs per self report; and
* female subjects of childbearing potential will be required to practice acceptable methods of birth control (the acceptable methods of birth control include birth control pills, Birth Control Shot, Birth Control Implant, IUD, Diaphragm, and cervical cap).
* if a participant takes kava dietary supplement, a 2-week washout period is needed for the participant to initiate this study or if a participant participated in a kava trial before, such as the kava JEK trial, the participant could be enrolled if the inclusion criteria above are met, including the 2-week washout period.

Exclusion Criteria:

* history of active cancer (other than non-melanoma skin cancer) within the past 2 years;
* diagnosed with liver dysfunction or with previous liver diseases;
* levels of alanine transaminase, aspartate transaminase, alkaline phosphatase or total bilirubin over limit of normal (ULN) range at prescreen;
* inability to refrain from acetaminophen, alcohol (no more than one drink daily via self-report), or other potentially hepatotoxic substances;
* are pregnant or nursing (lactating) or of childbearing age planning to become pregnant or unwilling to use adequate contraception during the study;
* participant answered "Yes" to any of the Modified Ask Suicide Screening Questions questions 1 through 3, or refuses to answer all of the questions. If subject answers 'Yes' to question 4 but the most recent suicide attempt took place >12 months from screening visit then subject is still eligible.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Subject Compliance with Intervention | 4 weeks
  Evaluate subject compliance with the kava intervention, as measured by participant reported number of missed doses
Subject Compliance with Intervention | 4 weeks
  Evaluate subject compliance with the kava intervention, as measured by detection of dihydromethysticin in participant urine by urine testing

SECONDARY OUTCOMES:
Tobacco cessation | 12 weeks
  Examine whether kava has the potential to help facilitate tobacco cessation, as measured by participant reported number of cigarettes smoked
Tobacco cessation | 12 weeks
  Examine whether kava has the potential to help facilitate tobacco cessation, as measured by the Fagerström Test for Nicotine Dependence (FTND)
Tobacco cessation | 12 weeks
  Examine whether kava has the potential to help facilitate tobacco cessation, as measured by the Modified Cigarette Evaluation Questionnaire (mCEQ)
Tobacco cessation | 12 weeks
  Examine whether kava has the potential to help facilitate tobacco cessation, as measured by the Brief Questionnaire on Smoking Urges (QSU-Brief)
Tobacco cessation | 12 weeks
  Examine whether kava has the potential to help facilitate tobacco cessation, as measured by urinary total nicotine equivalents
Effect on stress | 12 weeks
  Examine whether kava has the potential to reduce stress, as measured by the Perceived Stress Scale (PSS). The Perceived Stress Scale consists of 10 items that are each scored on a scale of 0-4. The maximum possible score for this instrument is 40 and the minimum score is 0. A higher score indicates greater perceived stress.
Effect on stress | 12 weeks
  Examine whether kava has the potential to reduce stress, as measured by plasma PRKACA
Effect on stress | 12 weeks
  Examine whether kava has the potential to reduce stress, as measured by plasma cortisol
Effect on stress | 12 weeks
  Examine whether kava has the potential to reduce stress, as measured by urinary TCE
Effect on stress | 12 weeks
  Examine whether kava has the potential to reduce stress, as measured by total cortisol equivalents
Effect on sleep | 12 weeks
  Examine whether kava has the potential to improve sleep, as measured by the Insomnia Severity Scale. The Insomnia Severity Scale instrument consists of 7 items that are each scored on a scale of 0-4. The maximum possible score for this instrument is 28 and the minimum score is 0. A higher score indicates more severe insomnia.
Effect on sleep | 12 weeks
  Examine whether kava has the potential to improve sleep, as measured by the Pittsburgh Sleep Quality Index (PSQI)
Effect on sleep | 12 weeks
  Examine whether kava has the potential to improve sleep, as measured by urinary 6-hydroxymelatonin
Effect on sleep | 12 weeks
  Examine whether kava has the potential to improve sleep, as measured by urinary N-acetyl serotonin
Effect on sleep | 12 weeks
  Examine whether kava has the potential to improve sleep, as measured by urinary NAS

CONTACTS AND LOCATIONS:
Overall Officials: Ramzi Salloum, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Xing C, Malaty J, Malham MB, Orlando FA, Lynch A, Huo Z, Francois M, Firpi-Morell R, Fisher CL, Christou DD, Salloum RG. The potential of AB-free kava in enabling tobacco cessation via management of abstinence-related stress and insomnia: study protocol for a randomized clinical trial. BMC Complement Med Ther. 2024 Dec 21;24(1):422. doi: 10.1186/s12906-024-04722-9. PMID 39709468

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT05814055/Prot_SAP_000.pdf